CLINICAL TRIAL: NCT04559204
Title: A Multi-centered, Randomized, Controlled Study to Evaluate the Safety and Immunogenicity of Combined Immunization of 23-valent Pneumococcal Polysaccharide Vaccine (PPV23) and Quadrivalent Inactivated Influenza Vaccine (IIV4)
Brief Title: Evaluation of Safety and Immunogenicity of Combined Immunization of PPV23 and IIV4
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: China National Biotec Group Company Limited (Industry)
Collaborators: Center for Disease Control and Prevention, Fujian (Other); Chengdu Institute of Biological Products Co.,Ltd. (Industry); Changchun Institute of Biological Products Co., Ltd. (Industry); National Institutes for Food and Drug Control, China (Other); Guizhou Center for Disease Control and Prevention (Other); Hunan Provincial Center for Disease Control and Prevention (Other); Peking University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IIV4-PPV23
Record Dates: First submitted 2020-09-09; First posted 2020-09-22 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-08

CONDITIONS: Influenza, Human; Pneumonia, Pneumococcal
Keywords: 23-valent Pneumococcal Polysaccharide Vaccine; Quadrivalent Inactivated Influenza Vaccine
MeSH Terms: conditions — Influenza, Human; Pneumonia, Pneumococcal

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- experimental group (Experimental): 408 subjects from experimental group will be simultaneously administrated with one dose of IIV (0.5 ml) and one dose of PPV23 (0.5 ml). Blood samples are collected before vaccination and one month (30 days) later.
  Interventions: Biological: IIV4 and PPV23
- control group A (Active Comparator): 408 subjects from control group A will be only administrated with one dose of IIV (0.5 ml). Blood samples are collected before vaccination and one month (30 days) later.
  Interventions: Biological: IIV4
- control group B (Active Comparator): 408 subjects from control group B will be only administrated with one dose of PPV23 (0.5 ml). Blood samples are collected before vaccination and one month (30 days) later.
  Interventions: Biological: PPV23

INTERVENTIONS:
Biological: IIV4 and PPV23 — imultaneously immunization of 23-valent pneumococcal polysaccharide vaccine (PPV23) and quadrivalent inactivated influenza vaccine (IIV4)
  Arms: experimental group
Biological: IIV4 — administrated with IIV4 only
  Arms: control group A
Biological: PPV23 — administrated with PPV23 only
  Arms: control group B

SUMMARY:
Subjects will be recruited and divided into 3 groups:

1. Experimental Group (408 subjects): combined immunization of PPV23 and IIV4;
2. Control Group A (408 subjects): IIV4 only;
3. Control Group B (408 subjects): PPV23 only;

All blood samples will be collected before and one month after vaccinatioin. The immunogenicity and safety of both experimental and control groups will be compared and the data be analyzed.

DETAILED DESCRIPTION:
To evaluate the safety and immunogenicity of simultaneously immunization of 23-valent pneumococcal polysaccharide vaccine (PPV23) and quadrivalent inactivated influenza vaccine (IIV4) , we design this randomized, parallel controlled study . 1224 subjects are divided into 3 groups, including 1 experimental group and 2 control groups (control group A and B), each group includes 408 subjects respectively.

Each 408-subject group is divided again into 4 age-based subgroups: ① 3-8 years old; ② 9-18 years old; ③ 19-49 years old ; ④ over 50 years old; each subgroup includes 102 subjects respectively.

408 subjects from experimental group will be simultaneously administrated with one dose of IIV (0.5 ml) and one dose of PPV23 (0.5 ml). Blood samples are collected before vaccination and one month (30 days) later.

408 subjects from control group A will be only administrated with one dose of IIV (0.5 ml). Blood samples are collected before vaccination and one month (30 days) later.

408 subjects from control group B will be only administrated with one dose of PPV23 (0.5 ml). Blood samples are collected before vaccination and one month (30 days) later.

To evaluate the immunogenicity, we will detect and compare the neutralization antibody levels, the seroprotection rates, and antibody geometric mean concentrations. The safety of all groups will be monitored as well.

ELIGIBILITY:
Inclusion Criteria:

* subjects aged no younger than 3 years old on the day of recruitment;
* with valid informed consent signed by parent(s) or guardian(s);
* parent(s) or guardian(s) are able to attend all scheduled appointments and comply with all study instructions;
* subjects have not received any seasonal influenza vaccine or pneumonia vaccine before;
* axillary temperature ≤37.0℃

Exclusion Criteria:

* subject who has a medical history with hypersensitiveness, eclampsia, epilepsy, cerebropathia or neurological illness;
* allergic to any ingredient of vaccine or with allergy history to any vaccine;
* subjects with immunodeficency or suspected impairment of immunologic function (e.g. caused by HIV), or subjects are in the process of immunosuppressor therapy(taking orally injecting of steroid hormone);
* administration of immunoglobulins within 30 days prior to this study;
* acute febrile disease(temperature ≥ 37.0°C) or infectious disease;
* have a clearly diagnosed history of thrombocytopenia or other coagulopathy, which might cause contraindications for subcutaneous injection;
* any serious chronic illness, acute infectious diseases, or respiratory diseases; severe cardiovascular disease, liver and kidney diseases or diabetes mellitus with complications;
* any kind of infectious, purulent, or allergic skin diseases;
* pregnant women and breastfeeding women;
* inoculated with any vaccine within 14 days of the study;
* any other factor that makes the investigator determines the subject is unsuitable for this study.

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1224 (Actual)
Dates: Start 2020-09-11 (Actual); Primary Completion 2020-11-26 (Actual); Study Completion 2021-10-09 (Actual)

PRIMARY OUTCOMES:
Seroconversion rate (IIV4) | Baseline (before vaccination) results
  the rate of positive seroconversion against influenza A (H3N2, H1N1) type and B (BY, BV) type viruses
Seroconversion rate (IIV4) | Results obtained 1 month after vaccination
  the rate of positive seroconversion against influenza A (H3N2, H1N1) type and B (BY, BV) type viruses
Seroconversion rate (PPV23) | Baseline (before vaccination) results
  the rate of positive seroconversion against 23 pneumococcal serotypes
Seroconversion rate (PPV23) | Results obtained 1 month after vaccination
  the rate of positive seroconversion against 23 pneumococcal serotypes
Geometric Mean Concentration (GMC) (IIV4) | Baseline (before vaccination) results
  GMCs of influenza A (H3N2, H1N1) type and B (BY, BV) type viruses
Geometric Mean Concentration (GMC) (IIV4) | Results obtained 1 month after vaccination
  GMCs of influenza A (H3N2, H1N1) type and B (BY, BV) type viruses
Geometric Mean Concentration (GMC) (PPV23) | Baseline (before vaccination) results
  GMCs of 23 pneumococcal serotypes
Geometric Mean Concentration (GMC) (PPV23) | Results obtained 1 month after vaccination
  GMCs of 23 pneumococcal serotypes

SECONDARY OUTCOMES:
adverse events following vaccination | 0-1 month (30 days)
  analyse the incidence of adverse events following immunization, both solicited and unsolicited

CONTACTS AND LOCATIONS:
Overall Officials: Shanying Zhang, Principal Investigator — Center for Disease Control and Prevention, Fujian
Locations (4):
- China (4):
  - Liucheng Community Health Services Center, Quanzhou, Fujian
  - Luodong County Health Center, Quanzhou, Fujian
  - Qingzhen Center for Disease Control and Prevention, Qingzhen, Guizhou
  - Qidong County Center for Disease Control and Prevention, Hongqiao, Hunan

IPD SHARING:
Plan to Share IPD: No